CLINICAL TRIAL: NCT06165939
Title: Effectiveness of Hydrodilatation With Hypertonic Dextrose Solution Injection After Intra-articular Steroid Injection for Frozen Shoulder Treatment: A Randomized Controlled Trial
Brief Title: Hydrodilatation With Hypertonic Dextrose Solution Injection After Intra-articular Steroid Injection for Frozen Shoulder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, Chih-Ya Chang, Doctor, Tri-Service General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: B202305141
Record Dates: First submitted 2023-12-03; First posted 2023-12-12 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Frozen Shoulder
Keywords: Frozen Shoulder; hypertonic dextrose injection; Steroid Injection; Hydrodilatation
MeSH Terms: conditions — Bursitis | interventions — Adrenal Cortex Hormones; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intra-articular corticosteroid injection and hydrodilation with 15% hypertonic dextrose (Experimental): The patient receives ultrasound-guided intra-articular corticosteroid injection treatment in the shoulder joint (2 ml SHINCORT INJ 10 MG/ML + 2 ml 2% Xylocaine). Subsequent assessments occur at the second and fourth weeks, followed by a second round of ultrasound-guided shoulder joint injection with 15% hypertonic dextrose (6 ml 50% Dextrose + 2 ml 2% Xylocaine + 12 ml Normal saline, totaling 20 ml). The entire treatment comprises two sessions.
  Interventions: Drug: Intra-articular corticosteroid injection; Drug: hydrodilation with 15% hypertonic dextrose
- Intra-articular corticosteroid injection and hydrodilation with Normal saline (Placebo Comparator): The patient receives ultrasound-guided intra-articular corticosteroid injection treatment in the shoulder joint (2 ml SHINCORT INJ 10 MG/ML + 2 ml 2% Xylocaine). Subsequent assessments occur at the second and fourth weeks, followed by a second round of ultrasound-guided shoulder joint injection with 15% hypertonic dextrose ( 2 ml 2% Xylocaine + 18 ml Normal saline, totaling 20 ml). The entire treatment comprises two sessions.
  Interventions: Drug: Intra-articular corticosteroid injection; Drug: hydrodilation with Normal saline

INTERVENTIONS:
Drug: Intra-articular corticosteroid injection — Ultrasound-guided intra-articular corticosteroid injection treatment in the shoulder joint (2 ml SHINCORT INJ 10 MG/ML + 2 ml 2% Xylocaine) is performed once for the patient at the first week.
Drug: hydrodilation with 15% hypertonic dextrose — The second round of ultrasound-guided shoulder joint injection is performed at the fourth week during the follow-up period and the injectate is 15% hypertonic dextrose (6 ml 50% Dextrose + 2 ml 2% Xylocaine + 12 ml normal saline, totaling 20 ml).
  Arms: Intra-articular corticosteroid injection and hydrodilation with 15% hypertonic dextrose
Drug: hydrodilation with Normal saline — The second round of ultrasound-guided shoulder joint injection is performed at the fourth week during the follow-up period and the injectate is Normal saline (2 ml 2% Xylocaine + 18 ml normal saline, totaling 20 ml).
  Arms: Intra-articular corticosteroid injection and hydrodilation with Normal saline

SUMMARY:
This study aims to investigate whether intra-articular corticosteroid injection, followed by hypertonic dextrose injection and shoulder joint capsular distension, is more effective than saline injection and shoulder joint capsular distension for treating frozen shoulder.

DETAILED DESCRIPTION:
Frozen shoulder (FS), also known as adhesive capsulitis, is a prevalent shoulder condition, with an annual incidence of around 2.4 individuals per 100,000, representing approximately 2% of the total population. Symptoms typically manifest in individuals aged forty to sixty years, characterized by persistent limitations in shoulder joint mobility accompanied by pain.

While the specific mechanisms driving frozen shoulder remain unclear, arthroscopic examination of the shoulder joint reveals thickening and contraction of the shoulder joint capsule, adhesion with the humeral head, and a reduction in joint cavity volume, particularly in the folds of the axillary recess of the joint capsule and its surrounding areas. These changes contribute to restricted shoulder joint mobility. Additionally, research suggests that severe inflammation may lead certain cytokines and growth factors to drive fibroblasts to replace normal tissue through repair and remodeling responses. This excessive fibrosis, along with the loss of a normal collagen remodeling response, further contributes to the development of frozen shoulder.

The 2020 meta-analysis published in JAMA Network underscored the importance of medium to long-term physical therapy in enhancing subsequent improvements in range of motion and functionality for patients with adhesive capsulitis or frozen shoulder. Furthermore, numerous studies indicate that combining intra-articular injections with shoulder joint capsular distension procedures, such as hydrodilatation, can enhance shoulder joint function and mobility.

Prolotherapy, a non-surgical regenerative injection therapy, involves injecting a solution into painful or degenerated areas. The injected proliferants induce a local inflammatory response, triggering the release of growth factors and stimulating fibroblasts and collagen-producing cells. This process mimics the natural healing mechanisms of the body, promoting cellular tissue growth through a beneficial inflammatory response. In clinical practice, the most commonly utilized solution for prolotherapy is hypertonic dextrose, with concentrations ranging from 15% to 25%. Concentrations exceeding 10% are generally considered to induce local inflammation, thereby initiating a cascade of reparative effects.

Although numerous studies have investigated shoulder joint capsular distension procedures in the past, the injected solutions often comprised corticosteroids and saline. In clinical observations, the use of hypertonic dextrose injection combined with shoulder joint capsular distension appears to yield improved outcomes in terms of pain relief and joint angle progression in patients with adhesive capsulitis. However, there is currently no research investigating the effectiveness of hypertonic dextrose injection combined with shoulder joint capsular distension for treating frozen shoulder. This study aims to explore whether intra-articular corticosteroid injection, followed by hypertonic dextrose injection and shoulder joint capsular distension, is more effective than saline injection and shoulder joint capsular distension for treating frozen shoulder.

ELIGIBILITY:
Inclusion Criteria:

1. The diagnosis of frozen shoulder is determined by physicians through an evaluation of the patient's medical history, physical examination, and assessment of X-ray and ultrasound reports.
2. The duration of symptoms should be more than 3 months.
3. There should be a decrease of at least 30 degrees in a minimum of two shoulder joint angles (shoulder flexion, abduction, and external rotation) compared to the corresponding angles on the healthy side.

Exclusion Criteria:

1. Ultrasound examination of the shoulder muscles must not reveal a complete tear or massive tear of the rotator cuff tendon or evidence of calcific tendinitis.
2. Presence of systemic rheumatic disease.
3. History of previous shoulder fracture or undergoing surgical intervention.
4. Receipt of shoulder joint injections within the last 3 months.
5. Acute cervical nerve root compression.
6. Current status of pregnancy or breastfeeding.
7. Poorly controlled diabetes (since intravenous glucose injection may cause temporary blood sugar elevation).
8. Patients with a history of cancer.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | the change from baseline, post-intervention 2, 4, 8, 12 weeks and 6 months
  The visual analogue scale (VAS) is a scale used to determine the pain intensity experienced by individuals. "0" means painless and "10" means extremely painful.

SECONDARY OUTCOMES:
Range of Motion (ROM) | the change from baseline, post-intervention 2, 4, 8, 12 weeks and 6 months
  Using a standardized goniometer, passive shoulder joint range of motion angles on the affected side are measured in standard positions, including flexion, extension, abduction, external rotation, and internal rotation.
Shoulder Pain and Disability Index (SPADI) | the change from baseline, post-intervention 2, 4, 8, 12 weeks and 6 months
  Shoulder function and disability were evaluated using the Chinese version of the Shoulder Pain and Disability Index (SPADI), a self-report questionnaire that yields pain and disability domain and total scores. The SPADI includes five questions on pain and eight questions on disability, referring to various problems with the shoulder encountered over the preceding week. Each item's score ranges from 0 (no pain/normal) to 10 (maximal pain/disability), with total scores of pain from 0-50 and disability from to 0-80. A higher score shows more disability.